CLINICAL TRIAL: NCT05936801
Title: Comparative Effects of Anterior Chest Compression Assist and Abdominal Thrust Assist Technique on Sputum Diary, Oxygen Saturation, Expiratory Flow Rate, and Dyspnea in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Comparison of Anterior Chest Compression Assist and Abdominal Thrust Assist Technique COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0323
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A total 34 patients will be taken. 2 groups will be created to apply intervention. After signing consent form, 17 patients in group A will be given abdominal thrust assist technique and 17 patients in group B will be given anterior chest compression technique. Baseline treatment given to both groups will include percussion and tapping.
Who Masked: Participant
Masking Description: A total 34 patients will be taken. 2 groups will be created to apply intervention. After signing consent form, 17 patients in group A will be given abdominal thrust assist technique and 17 patients in group B will be given anterior chest compression technique. Baseline treatment given to both groups will include percussion and tapping. The data collected will then be analyzed using IBM SPSS version 25
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Chest Compression technique (Experimental): Baseline treatment given is percussion and vibration in side lying position. The therapist puts one arm across the patient's pectoral region to stabilize or compress the upper chest while the other arm is placed either parallel on the lower chest or abdomen below the xiphoid process. Inspiration is facilitated by the pressure on anterior chest, followed by a "hold."
  Just as the patient is instructed to cough, the therapist applies a quick force with both arms:
  down and back on the upper chest and up and back on the lower chest or abdomen. 3 sessions in a wk would be given on alternate days
  Interventions: Other: Anterior Chest Compression technique
- Abdominal Thrust Technique (Experimental): Baseline treatment given is percussion and vibration in side lying position. It Can be used in both the supine and side lying positions. With the patient in the supine position, the therapist places the heel of one hand inferior to the patient's xiphoid process and below the patient's lower ribs.
  Interventions: Other: Abdominal Thrust Technique

INTERVENTIONS:
Other: Anterior Chest Compression technique — Baseline treatment given is percussion and vibration in side lying position. The therapist puts one arm across the patient's pectoral region to stabilize or compress the upper chest while the other arm is placed either parallel on the lower chest or abdomen below the xiphoid process. Inspiration is facilitated by the pressure on anterior chest, followed by a "hold."
  Just as the patient is instructed to cough, the therapist applies a quick force with both arms:
  down and back on the upper chest and up and back on the lower chest or abdomen. 3 sessions in a wk would be given on alternate days Baseline treatment given is percussion and vibration in side lying position. It Can be used in both the supine and side lying positions. With the patient in the supine position, the therapist places the heel of one hand inferior to the patient's xiphoid process and below the patient's lower ribs.
  Other Names: Abdominal Thrust Technique
  Arms: Anterior Chest Compression technique
Other: Abdominal Thrust Technique — Baseline treatment given is percussion and vibration in side lying position. It Can be used in both the supine and side lying positions. With the patient in the supine position, the therapist places the heel of one hand inferior to the patient's xiphoid process and below the patient's lower ribs.
  Arms: Abdominal Thrust Technique

SUMMARY:
A total 34 patients will be taken. 2 groups will be created to apply intervention. After signing consent form, 17 patients in group A will be given abdominal thrust assist technique and 17 patients in group B will be given anterior chest compression technique.

DETAILED DESCRIPTION:
Patient is instructed to take in a deep breath and hold it. Then, just as the patient is instructed to cough, the therapist applies a quick push up and in under the diaphragm with the heel of the hand. In Anterior chest compression: the therapist places one arm across the patient's pectorals and the other parallel to it. After the patient takes a maximal breath, the therapist pushes down to help the patient cough. The greatest force is applied through the lower chest during expulsion. A total 34 patients will be taken. 2 groups will be created to apply intervention. After signing consent form, 17 patients in group A will be given abdominal thrust assist technique and 17 patients in group B will be given anterior chest compression technique. Baseline treatment given to both groups will include percussion and tapping. The data collected will then be analyzed using IBM SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* uncontrolled Tachycardia
* Unconscious patients
* In neuro-compromised patients with Cognitive dysfunction
* Recent esophageal surgery
* Acute abdominal distension -Recent Broncho-pleural fistula - Pulmonary embolism, pneumothorax hemothorax
* Unstable head and neck fracture

Exclusion Criteria:

* Breathlessness, Cough and sputum scale (BCSS)
* Modified Borg Dyspnea scale
* Peak Flow Meter
* Pulse Oximeter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
sputum diary | 4 weeks
  sputum of each patient will be recorded.
Oxygen saturation | 4 weeks
  oxygen saturation will be measure with pulse oximeter.
expiratory flow rate | 4 weeks
  Expiratory flow rate will be measured through peak expiratory flow meter

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital, Rahim Yar Khan., Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petty TL. The history of COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(1):3-14. doi: 10.2147/copd.2006.1.1.3. PMID 18046898
- [Background] Lopez-Campos JL, Calero C, Quintana-Gallego E. Symptom variability in COPD: a narrative review. Int J Chron Obstruct Pulmon Dis. 2013;8:231-8. doi: 10.2147/COPD.S42866. Epub 2013 May 7. PMID 23687444
- [Background] Ramos FL, Krahnke JS, Kim V. Clinical issues of mucus accumulation in COPD. Int J Chron Obstruct Pulmon Dis. 2014 Jan 24;9:139-50. doi: 10.2147/COPD.S38938. eCollection 2014. PMID 24493923
- [Background] Liao LY, Chen KM, Chung WS, Chien JY. Efficacy of a respiratory rehabilitation exercise training package in hospitalized elderly patients with acute exacerbation of COPD: a randomized control trial. Int J Chron Obstruct Pulmon Dis. 2015 Aug 27;10:1703-9. doi: 10.2147/COPD.S90673. eCollection 2015. PMID 26345529
- [Background] Andersen TM, Hov B, Halvorsen T, Roksund OD, Vollsaeter M. Upper Airway Assessment and Responses During Mechanically Assisted Cough. Respir Care. 2021 Jul;66(7):1196-1213. doi: 10.4187/respcare.08960. Epub 2021 Feb 12. PMID 33579747
- [Background] Hughes R, Rapsomaniki E, Janson C, Keen C, Make BJ, Burgel PR, Tomaszewski EL, Mullerova H, Reddel HK; NOVELTY study investigators. Frequent productive cough: Symptom burden and future exacerbation risk among patients with asthma and/or COPD in the NOVELTY study. Respir Med. 2022 Aug-Sep;200:106921. doi: 10.1016/j.rmed.2022.106921. Epub 2022 Jun 20. PMID 35820227